CLINICAL TRIAL: NCT05026697
Title: Validity and Reliability of Commercially Available Bioelectrical Impedance Analysis Devices
Acronym: CBIA
Status: Completed | Type: Observational
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB2021-107
Record Dates: First submitted 2021-06-03; First posted 2021-08-30 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Body Composition
Keywords: body composition; fat mass; fat-free mass; body fat percentage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this data collection is to establish the validity and reliability of several different commercially available bioelectrical impedance analysis devices that are used to estimate body composition.

DETAILED DESCRIPTION:
The purpose of this data collection is to establish the validity and reliability of several different commercially available bioelectrical impedance analysis devices that are used to estimate body composition.

This study will involve 1-2 total visits: one initial visit followed by an optional follow-up visit 12-16 weeks later. These visits will consist of body composition assessments after an overnight fast. Before the overnight fast, the individual will be asked to drink 1 liter (the equivalent of two 16.9-ounce water bottles) between the final meal of the day and the beginning of the 8-hour fasting period. At the first visit, participants will undergo dual x-ray absorptiometry (DXA; GE Lunar Prodigy), air displacement plethysmography (ADP; Cosmed Bod Pod), a 3D body scan (SizeStream SS20), and several multi- and single-frequency bioelectrical impedance analysis (BIA) assessments. The BIA assessment methods will be conducted twice. This will allow for test-retest reliability assessment of each of the BIA devices being assessed in our study. At the optional second visit, all assessment methods utilized in our laboratory will be conducted once. By comparing these values to the values from the first visit, we will be able to establish the cumulative error due to technical error and biological error (i.e. random biological differences in the participants between the two assessments). We will collect data in a similar fashion during this second visit in order to compare the changes over time between the measurements provided by the commercially available BIA devices against the changes detected by a validated 4-compartment model of body composition, which uses research-grade devices. Cumulatively, this information will provide essential data to consumers regarding both the immediate and long-term test-retest reliability as well as the validity of commercially available BIA devices such as home body fat scales.

The commercially available BIA devices being examined in the present study includes:

* Omron HBF-306
* RENPHO Smart Bathroom Scale (item number: ES-26BB-B)
* Hawanna Body Fat Scale (UPC: 791555289926)
* Wyze Scale (SKU: WHSCL1)
* INEVIFIT Smart Body Fat Scale (UPC: 711841680565; EAN: 0711841680565)
* WeightWatchers Scale by Conair (model: WW721XF)
* Tanita UM-081 (model: UM-081; EAN: 0742496801012 and 0885157966993)
* VitaGoods FormFit Digital Scale and Body Analyzer (model: VG42252-0000)
* Omron HBF 516 Body Composition Monitor (model: HBF-516B)
* Seca sensa 804
* Withings/Nokia BodyCardio Body Composition Digital Scale (model: WBS04b-Black-All-Inter)
* Tanita BC554 IronMan Body Composition Monitor (model: BC-554)
* Tanita BC568 InnerScan Segmental Body Composition Monitor (model: BC-568)
* InBody H2ON Smart Full Body Composition Analyzer

Additionally, several laboratory-grade bioimpedance technologies will be performed, including ImpediMed SFB7 bioimpedance spectroscopy and Seca mBCA 515/514 multi-frequency bioelectrical impedance analysis. Urine specific gravity will also be assessed using digital refractometry, and height will be assessed via stadiometer. As part of the ADP test, body mass estimates from a calibrated, research-grade scale will be obtained (Modified BWB-627-A, Tanita Corporation).

The test-retest reliability of the commercially available bioelectrical impedance analysis devices will be examined through duplicate assessments. The validity of the commercially available bioelectrical impedance analysis devices will be examined as compared to the criterion laboratory methods, namely the 4-compartment model for total body composition and DXA and/or laboratory-grade segmental bioimpedance technologies for segmental body composition.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50
* Generally healthy (defined as an absence of any disease or medical condition which could potentially result in abnormal body composition, including but not limited to musculoskeletal or metabolic diseases)
* Weight-stable (defined as no change in body mass >5 pounds in the past month)

Exclusion Criteria:

* Failing to meet any of the aforementioned inclusion criteria or self-reporting a body composition abnormality (due to medical condition, lifestyle practices, etc.)
* Height greater than 75.5 inches (due to height limitation of DXA scanner)
* Weight greater than 330 pounds (due to weight limitation of some of the devices used)
* Presence of facial hair longer than 1/2 inch (and unwillingness to shave) or self-report of large amounts of body hair due to the impact of hair on Bod Pod body volume estimates
* Presence of pacemaker or any electrical device (due to electrical currents administered by bioimpedance devices)
* Amputation of limb, implantation of a meaningful amount metal (e.g., full joint replacement), or physical deformity large enough to invalidate traditional body composition assessments

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of generally healthy, weight-stable adults located in or near the community of Lubbock, Texas (or willing to travel to Lubbock, Texas).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Body fat percentage | 1 day
  Percentage of body mass that is attributable to fat mass. This value is provided by each body composition assessment device being tested (see list of devices in Study Description).
Fat-free mass | 1 day
  Calculated as body mass minus fat mass. Fat mass is equal to body mass multiplied by body fat percentage. Body fat percentage is provided by each body composition assessment device being tested (see list of devices in Study Description).
Fat mass | 1 day
  Body mass multiplied by body fat percentage. Body fat percentage is provided by each body composition assessment device being tested (see list of devices in Study Description).

SECONDARY OUTCOMES:
Segmental body fat percentage | 1 day
  Body fat percentage provided for specific body segments (i.e., trunk/torso, arms, and legs). These values are provided by some, but not all, of the body composition assessment devices being tested (see list of devices in Study Description).
Segmental fat-free mass | 1 day
  Fat-free mass (i.e., body mass minus fat mass) provided for specific body segments (i.e., trunk/torso, arms, and legs). These values are provided by some, but not all, of the body composition assessment devices being tested (see list of devices in Study Description).
Segmental fat mass | 1 day
  Fat mass provided for specific body segments (i.e., trunk/torso, arms, and legs). These values are provided by some, but not all, of the body composition assessment devices being tested (see list of devices in Study Description).

OTHER OUTCOMES:
Body mass | 1 day
  Body mass estimates provided by the scale of each body composition assessment device (see list of devices in Study Description).
Total body water | 1 day
  Mass of total body water. These values are provided by some, but not all, of the body composition assessment devices being tested (see list of devices in Study Description).
Visceral fat | 1 day
  Mass of visceral fat. These values are provided by some, but not all, of the body composition assessment devices being tested (see list of devices in Study Description).
Bone mineral mass | 1 day
  Mass of bone mineral; These values are provided by some, but not all, of the body composition assessment devices being tested (see list of devices in Study Description).

CONTACTS AND LOCATIONS:
Overall Officials: Grant Tinsley, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided